CLINICAL TRIAL: NCT02219672
Title: Study on the Impact of Triptolide Woldifiion on HIV-1 Reservoir of Chinese HIV/AIDS Patients In Acute HIV-1 Infection
Brief Title: Study on the Impact of Triptolide Woldifiion on HIV-1 Reservoir In Acute HIV-1 Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, LI Taisheng, department of the infectious disease, Peking Union Medical College
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CACT140816
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: AIDS/HIV PROBLEM
Keywords: Triptolide wilfordii HIV-1 reservoir acute hiv infection
MeSH Terms: interventions — Tenofovir; Lamivudine; Lopinavir; Ritonavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptolide group (Experimental): cART for 6 months, and the experimental group will take Triplitode 2 tabs tid po for another 12 months
  Interventions: Drug: Triplitode
- Comparator group (Active Comparator): combined antiretroviral therapy (cART): TDF+3TC+LPV/r+RAL for 18 months
  Interventions: Drug: Tenofovir plus lamivudine plus Lopinavir / ritonavir plus raltegravir

INTERVENTIONS:
Drug: Triplitode — Drug: Triptolide Triptolide Wilfordii is a Chinese old herb which is widely used as a remedy for rheumatic diseases and nephropathy in China. It is approved that it can play a role as an immune modular.
  Other Name: Tripterygium Wilfordii Hook F (TwHF) Drug: cART Participants who will be enrolled in this Triplitode group would be treated with Tenofovir plus lamivudine plus Lopinavir / ritonavir plus raltegravir .
  Other Names: Triptolide Wilfordii
  Arms: Triptolide group
Drug: Tenofovir plus lamivudine plus Lopinavir / ritonavir plus raltegravir — Participants who will be enrolled in this trial would be treated with Tenofovir plus lamivudine plus Lopinavir / ritonavir plus raltegravir.
  Other Names: TDF+3TC+LPV/r+RAL for 18 months
  Arms: Comparator group

SUMMARY:
This study is a prospective trial which will recruit 18 patients in acute HIV-1 infection phase. This study aims to evaluate the effects and side effects of ARV treatment in Chinese patients in acute HIV-1 infection phase, and to evaluate the impact of Triptolide wilfordii on HIV-1 reservoir.

DETAILED DESCRIPTION:
Two arms will be enrolled in this study, 18 naive-treatment Chinese patients in acute HIV-1 infection phase would be allocated to two arms, and treated with the antiretroviral drugs (Tenofovir plus lamivudine plus Lopinavir / ritonavir plus raltegravir). Six months later, 12 patients will be treated with Triplitode, in order to observe the impact of of Triptolide wilfordii on HIV-1 reservoir of patients in acute infection phase. All patients should be explored for 18 months in terms of the clinical features, drugs side-effects, and immunological and viral response, and the HIV-1 reservoir. We hypothesis that Triptolide wilfordii might further reduce the HIV-1 reservoir. The result would provide proofs for further practical antiviral therapy for patients in acute infection phase in China or other resource limited countries.

ELIGIBILITY:
Inclusion Criteria:

* • age between 18-65 years

  * HIV seropositive and confirmed by western blot, confirmed as acute HIV-1 infection
  * good adherence and follow up in the same place
  * Inform Consent signed
  * ART-naïve

Exclusion Criteria:

* Active opportunistic infection (not stable within 4 weeks 2 weeks ) or AIDS-related carcinoma;

  * hemoglobin (HGB) < 9 g/dl 、 white blood cell (WBC) < 2000/ul 、 granulin (GRN) < 1000 /ul 、 platelet (PLT) < 75000 /ul 、 Cr >1.5x ULN 、 ALT or AST or alkaline phosphatase (ALP) >3x upper limit of normal (ULN) 、 total bilirubin (TBIL) >2x ULN 、 creatine kinase (CK) > 2x ULN;
  * Pregnant or breastfeeding woman or woman with pregnancy plan;
  * Active drug-user;Severe neurological defects;
  * Active alcohol abuse;
  * Severe gastrointestinal ulcer .
  * End-stage disease such as cirrhosis, chronic obstructive pulmonary disease, congestive heart failure, recent myocardial ischemia,tumor, etc
  * Those who are undertaking steroids, immunomodulator, anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Changes of the immunologic response, virologic response, and hiv-1 reservoir | baseline and at Week 4, Week 12, Week 24, Week 36 follow-up visits

SECONDARY OUTCOMES:
Adverse events of the therapy | thirty-six months

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China